CLINICAL TRIAL: NCT05359328
Title: RDS MultiSense® SpO2 Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhythm Diagnostic Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR 2022-466
Record Dates: First submitted 2022-04-25; First posted 2022-05-03 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2022-07

CONDITIONS: Hypoxia
Keywords: Hypoxia; Pulse Oximetry; SpO2; Remote Monitoring; Connected device; Real-time monitoring
MeSH Terms: conditions — Hypoxia | interventions — Respiratory Rate; Heart Rate; Vascular Access Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Controled Hypoxia - Healthy Volunteers (Other)
  Interventions: Device: Pulse Oximeter, Respiratory Rate, Heart Rate and Arterial line

INTERVENTIONS:
Device: Pulse Oximeter, Respiratory Rate, Heart Rate and Arterial line — Measurement of physiological parameters

SUMMARY:
The purpose of this clinical study is to validate the oxygen saturation (SpO2) accuracy of the RDS MultiSense® Pulse Oximetry during non-motion conditions over the range of 70-100% arterial oxygen saturation (SaO2) as compared to arterial blood samples assessed by measuring carbon monoxide (CO) bound to hemoglobin by CO-Oximetry. Additionally, data will be collected for heart rate accuracy as compared to reference ECG. The end goal is to provide supporting documentation for the SpO2 and heart rate accuracy validation for RDS MultiSense® Pulse Oximetry.

A minimum of 10 healthy adult male and female participants, ranging in age and pigmentation from light to dark, will be enrolled in the study to meet the study design requirements defined by International Organization for Standardization ISO 80601-2-61:2017: corrected version 2018-02 and by the FDA's Guidance for Pulse Oximeters (March 4, 2013). The participants will have an arterial catheter placed in the radial artery to allow for simultaneous blood samples during stable plateaus of induced hypoxic levels.

The investigational device will be placed on the placed on the thorax of the participants (patch on the upper back and external electrode on the right pectoral) per the instructions for use. Simultaneous data collection will be set up for the system under test and control oximeter.

ELIGIBILITY:
Inclusion Criteria:

* 10-15 Adults with a minimum of 3 males and a minimum of 3 females, with the balance made up of either
* Participant must have the ability to understand and provide written informed consent
* Participant is 18 to 50 years of age
* Participant must be willing and able to comply with study procedures and duration
* Participant is a non-smoker or who has not smoked within 2 days prior to the study

Exclusion Criteria:

* Participant is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, wrist, hands, ears or forehead/skull or other sensor sites, tattoo, extensive moles, or freckles in the optical path which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow participants to participate if the condition is noted and would not affect the particular sites utilized.)
* Female participants that are actively trying to get pregnant or are pregnant (confirmed by positive urine pregnancy test unless the participant is known to be not of child-bearing potential).
* Smoker participants who have refrained will be screened for Carboxyhemoglobin (COHb) levels >3% as assessed with a reference devie (Masimo Radical 7)
* Participants with known respiratory conditions (self-reported)
* Participants with known heart or cardiovascular conditions (self-reported, except for blood pressure and ECG review)
* Self-reported health conditions as identified in the Health Assessment Form (self-reported)
* Participants with known clotting disorders (self-reported)
* Participants with severe contact allergies to standard adhesives, silicon, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Participants with severe allergies to iodine (only applicable if iodine is used)
* Participants with severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocaine)
* Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test (Ratio < 0.4)
* Unwillingness or inability to remove colored nail polish from test digits.
* Unwillingness to have chest or other test sites shaved
* Other known health condition, should be considered upon disclosure in health assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Validation of SpO2 accuracy performance of RDS MultiSense® Pulse Oximeter by comparison to CO-Oximeter | From beginning to end of controled hypoxia, up to 2 hours
  The Accuracy Root Mean Square (Arms) value will be used as a metric. Reference CO-Oximetry will be used as the basis for comparison for the investigational device SpO2 readings.

SECONDARY OUTCOMES:
Evaluation of heart rate accuracy performance of RDS MultiSense® by comparison to ECG-derived heart rate | From beginning to end of monitoring, up to 2 hours
  The reference for comparison of the investigational device heart rate will be heart rate values collected from an ECG monitor.Heart rate accuracy will be assessed by review of the readings less than ±5 Beats Per Minute or ±10% from the Reference heart rate values.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimark LLC, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No